CLINICAL TRIAL: NCT02319668
Title: A Clinical Study to Evaluate the Efficacy of Pre-procedural and Pre-surgical Rinsing With an Antimicrobial Agent in Reducing Bacteria in Dental Aerosols and in the Oral Cavity
Brief Title: Antimicrobial Agent for Reducing Bacteria in Aerosols and Oral Cavity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202200; 2014-003222-40 (EudraCT Number); RH02604 (Other: GSK)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Dental Prophylaxis and Implant Surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test product (Experimental): Mouthwash containing 0.2% w/v Chlorhexidine digluconate
  Interventions: Drug: 0.2% w/v Chlorhexidine digluconate; Drug: Sodium fluoride toothpaste (Aquafresh Mild & Minty)
- Control (Placebo Comparator): Sodium fluoride toothpaste (Aquafresh Mild & Minty)
  Interventions: Drug: Sodium fluoride toothpaste (Aquafresh Mild & Minty)

INTERVENTIONS:
Drug: 0.2% w/v Chlorhexidine digluconate — Participants will brush their teeth with the reference product (toothpaste) and thoroughly rinse their mouth with water and wait 5 timed minutes before using 10 ml of the 0.2% w/v Chlorhexidine digluconate mouthwash, except when using at site, where no brushing will take place prior to using the mouthrinse.
  Arms: Test product
Drug: Sodium fluoride toothpaste (Aquafresh Mild & Minty) — Participants will apply a strip of toothpaste to cover the head of the toothbrush and will brush in their usual manner for two timed minutes twice daily. They will then rinse their mouth thoroughly with water after brushing

SUMMARY:
The primary objective of this study will be to evaluate the effect of two week pre-surgical rinsing with an antimicrobial mouthrinse containing 0.2% w/v Chlorhexidine digluconate on the total number of plaque bacteria in the mouth 3 days post implant surgery. The study will be conducted at Eastman Clinical Investigation Centre (ECIC), University College London (UCL) Eastman Dental Institute. Participants will be those who require a single and simple surgical implant to be placed, and will be recruited from new patient referrals within the Eastman Dental Hospital

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18-64 years old.
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general and mental health with, in the opinion of the investigator or medically qualified designee:

  1. No clinically significant and relevant abnormalities in medical history or upon oral examination.
  2. Absence of any condition that could affect the participant's safety or well being or their ability to understand and follow study procedures and requirements.
* Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception
* Dental Health

  1. Good overall oral health in the opinion of investigator.
  2. A minimum of 20 permanent teeth.
  3. Requiring a single and simple implant (single tooth replacement with no bone augmentation required for implant placement).
* Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Recent history (within the last 1 year) of alcohol or other substance abuse
* Use of antibiotics within 14 days prior to the Baseline visit or Implant surgery visit.
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the one center in the United kingdom.
Pre-assignment Details: A total of 44 participants were screened, out of which 38 were randomized. 6 participants were not randomized: 2 participants did not met study criteria, 2 participants withdrew their consent, 1 participant due to protocol violation, and 1 participant due to other reason (not specified).
Groups:
- Test and Reference Product: Participants rinsed for one timed minute with 10 milliliter (mL) of Test product (Mouthwash containing Chlorhexidine digluconate). Participants also applied a strip of reference product (toothpaste containing sodium fluoride) to cover the head of the toothbrush and brushed in their usual manner for two timed minutes first and thoroughly rinsed their mouth with water and waited for 5 timed minutes before using the mouthwash (except when used on site where they did not brush prior to using mouthwash).
- Reference Product: Participants applied a strip of reference product (toothpaste containing sodium fluoride) to cover the head of the toothbrush and brushed in their usual manner for two timed minutes. They then rinsed their mouth thoroughly with water after brushing.
Period: Overall Study
Arm/Group | Test and Reference Product | Reference Product
Started | 19 | 19
Completed | 19 | 17
Not Completed | 0 | 2
Not completed — Other (Not specified) | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population: defined as all the participants who were randomised and received at least one dose of study treatment during the study.
Groups:
- Test and Reference Product: Participants rinsed for one timed minute with 10 mL of Test product (Mouthwash containing Chlorhexidine digluconate). Participants also applied a strip of reference product (toothpaste containing sodium fluoride) to cover the head of the toothbrush and brushed in their usual manner for two timed minutes first and thoroughly rinsed their mouth with water and waited for 5 timed minutes before using the mouthwash (except when used on site where they did not brush prior to using mouthwash).
- Total: Total of all reporting groups
Arm/Group | Test and Reference Product | Reference Product | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (8.74) | 28.4 (12.23) | 27.9 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 18 | 14 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Detectable Plaque Bacteria Sampled 3 Days Post Implant Surgery
Description: The examiner identified three plaque sampling sites as follows: surgical site, contralateral site to the surgical site and tongue. An individual cotton swab was used at each identified site for up to 20 seconds in order to harvest a plaque sample and immediately be placed into 1mL phosphate buffered saline in a sterile Eppendorf tube. The samples were analysed using quantitative polymerase chain reaction (qPCR) which determined the total number of bacteria in a sample by quantifying the number of 16S ribosomal ribonucleic acid (rRNA) genes in the sample. The number of bacteria in each of the three identified plaque sampling sites (surgical site, contralateral site to the surgical site and tongue) for each participant were summed to calculate the total number of bacteria for each participant.
Time Frame: At Day 3
Population: Intent to treat (ITT) population (N=38): defined as all the participants who were randomised, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: log(10) colony forming equivalents (CFE)
Arm/Group | Test and Reference Product | Reference Product
Number analyzed (Participants) | 19 | 19
log(10) colony forming equivalents (CFE) | 7.63 (0.501) | 7.43 (0.598)
Statistical Analysis 1: Comparison: Test and Reference Product vs Reference Product; Test type: Superiority or Other; p = 0.2965, ANCOVA; ANCOVA with treatment as factor and baseline as covariate; Least square (LS) Mean difference = 0.20, 95% CI 2-sided [-0.18 to 0.58] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment

2. Secondary Outcome: Total Number of Detectable Plaque Bacteria Sampled at Implant Surgery (at Pre-rinse, Pre, Mid and Post Implant Surgery) and Post Implant Surgery (at Day 1 and 7)
Description: The examiner identified three plaque sampling sites as follows: surgical site, contralateral site to the surgical site and tongue. An individual cotton swab was used at each identified site for up to 20 seconds in order to harvest a plaque sample and immediately be placed into 1mL phosphate buffered saline in a sterile Eppendorf tube. The samples were analysed using quantitative polymerase chain reaction (qPCR) which determined the total number of bacteria in a sample by quantifying the number of 16S ribosomal ribonucleic acid (rRNA) genes in the sample.
Time Frame: At Day 0 (pre-rinse, pre, mid and post implant surgery), Day 1 and 7
Population: ITT (N=38) defined as all the participants who were randomised, received the study treatment at least once and provided at least one post-baseline assessment of efficacy. n was number of participants evaluated at specific endpoint.
Measure: Mean (Standard Deviation); unit: log (10) CFE
Groups:
- Test and Reference Products: Participants rinsed for one timed minute with 10 mL of Test product (Mouthwash containing Chlorhexidine digluconate). Participants also applied a strip of reference product (toothpaste containing sodium fluoride) to cover the head of the toothbrush and brushed in their usual manner for two timed minutes first and thoroughly rinsed their mouth with water and waited for 5 timed minutes before using the mouthwash (except when used on site where they did not brush prior to using mouthwash).
Arm/Group | Test and Reference Products | Reference Product
Number analyzed (Participants) | 19 | 19
log (10) CFE
  At Day 0 (pre rinse), (n=19,19) | 7.55 (0.376) | 7.74 (0.364)
  At Day 0 (pre implant), (n=19, 18) | 7.65 (0.375) | 8.01 (0.381)
  At Day 0 (mid implant), (n=19, 18) | 7.58 (0.449) | 7.84 (0.597)
  At Day 0 (post implant), (n=19,18) | 7.58 (0.429) | 7.81 (0.433)
  At Day 1 (n=19, 17) | 7.44 (0.409) | 7.06 (0.470)
  At Day 7 (n=19, 17) | 7.72 (0.335) | 7.38 (0.512)

3. Secondary Outcome: Area Under the Curve (AUC) for the Total Number of Plaque Bacteria in the Mouth Post Implant Surgery
Description: The examiner identified three plaque sampling sites as follows: surgical site, contralateral site to the surgical site and tongue. An individual cotton swab was used at each identified site for up to 20 seconds in order to harvest a plaque sample and immediately be placed into 1mL phosphate buffered saline in a sterile Eppendorf tube. The samples were analysed using quantitative polymerase chain reaction (qPCR) which determined the total number of bacteria in a sample by quantifying the number of 16S ribosomal ribonucleic acid (rRNA) genes in the sample. The AUC of the total count of detectable plaque bacteria was calculated using trapezoidal rule in the time range from immediately post implant surgery to 7 days post implant surgery
Time Frame: Up to 7 days post implant surgery
Population: ITT (N=38) defined as all the participants who were randomised, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: log (10) CFE × Day
Arm/Group | Test and Reference Product | Reference Product
Number analyzed (Participants) | 19 | 19
log (10) CFE × Day | 8.57 (0.319) | 8.37 (0.356)

4. Secondary Outcome: Total Number of Recoverable Viable Bacteria in the Aerosol Generated During Dental Prophylaxis
Description: Thick settle blood agar plates (supplemented with 5% [volume by volume v/v]) defibrinated horse blood) were used to determine the bacterial load of the aerosol. Thirty (30) minutes prior to the participants had their procedure (dental prophylaxis), a total of 5 settle plates with lids removed were placed at set positions around the dental surgery. After 30 minutes, the settle plates lids were replaced. This was repeated during the dental prophylaxis procedure using 5 fresh settle plates. All plates were then sealed with parafilm and transported for incubation in an anaerobic chamber at 37°C for 3 days. The plates were inspected daily to access growth and after 3 days removed and stored at 4°C for subsequent colony enumeration and Colony Forming Unit/mL (CFU/mL) calculation
Time Frame: At Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log (10) CFU/mL
Groups:
- Test and Reference Product: Participants rinsed for one timed minute with 10 mL of Test product only (mouthwash containing Chlorhexidine digluconate). Participants did not receive reference product(toothpaste containing sodium fluoride) during analysis of this outcome as this analysis was performed at baseline.
- Reference Product: Participants did not receive any product (mouthwash containing Chlorhexidine digluconate or toothpaste containing sodium fluoride) during analysis of this outcome as this analysis was performed at baseline.
Arm/Group | Test and Reference Product | Reference Product
Number analyzed (Participants) | 19 | 19
log (10) CFU/mL
  Pre prophylaxis | 0.94 (0.435) | 0.91 (0.606)
  Post prophylaxis | 1.31 (0.201) | 1.33 (0.326)

ADVERSE EVENTS:
Groups:
- Test and Reference Product: Participants rinsed for one timed minute with 10 mL of Test product (Mouthwash containing Chlorhexidine digluconate). Participants also applied a strip of reference product (toothpaste containing sodium fluoride) to cover the head of the toothbrush and brushed in their usual manner for two timed minutes first and thoroughly rinsed their mouth with water and waited for 5 timed minutes before using the mouthwash (except when used on site where they did not brushed prior to using mouthwash).
Arm/Group | Test and Reference Product | Reference Product
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 17/19 | 18/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test and Reference Product (N=19) | Reference Product (N=19)
Post procedural discomfort (Injury, poisoning and procedural complications) | 16 | 15
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 3
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 5 | 1
Ageusia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Tingue bitting (Nervous system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Lip exfoliation (Gastrointestinal disorders) | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0
Angular cheilitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Injury associated with device (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Implant site erythema (General disorders) | 0 | 2
Implant site haemorrhage (General disorders) | 0 | 1
Implant site pain (General disorders) | 0 | 1
Implant site swelling (General disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Urine ordour abnormal (Renal and urinary disorders) | 0 | 1
Oropharyngal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 3
Pain prophylaxis (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.